CLINICAL TRIAL: NCT03542760
Title: Use of Methylene Blue in Acquired Methemoglobinemia: Prospective Observational Registry (metHb)
Brief Title: Acquired Methemoglobinemia Observational Registry
Acronym: metHb
Status: Completed | Type: Observational
Sponsor: Hospital Quality Foundation (Other)
Collaborators: Prove pharm (Industry)
Responsible Party: Sponsor
Other Study IDs: HQF-METHB-2018001
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Methemoglobinemia, Acquired; Methemoglobinemia
Keywords: Methylene Blue
MeSH Terms: conditions — Methemoglobinemia | interventions — Methylene Blue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days

GROUPS / COHORTS (2):
- Primary Treated Group: Subjects who are administered methylene blue for treatment of acquired methemoglobinemia that is symptomatic (eg, exhibiting sleepiness, cyanosis, dizziness, etc) or with measured methemoglobin levels > 30%.
  Interventions: Drug: Methylene Blue
- Secondary Treated Group: Subjects who are administered methylene blue for treatment of acquired methemoglobinemia with measured methemoglobin levels ≤ 30 and lack of clinical symptoms
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Administration of methylene blue as per the treating physician's diagnosis and the acute care facility's standard of care

SUMMARY:
This prospective, observational registry aims to collect real-world data regarding the safety and efficacy of ProvayBlue® (methylene blue 0.5%) used according to normal standard of care for the treatment of acquired methemoglobinemia. Methylene blue has been used for decades as a rescue medication for the treatment of methemoglobinemia, a rare and potentially life-threatening condition in which elevated levels of methemoglobin impede the delivery of oxygen from blood to body tissues. However, consistent prospective data about the safety and efficacy of this medication are sparse, simply because of the rarity of the disorder. ProvayBlue® received accelerated FDA approval for treatment of acquired methemoglobinemia in 2016. This large, prospective, multi-center observational registry has been initiated to gain more information on the use of methylene blue in the treatment of acquired methemoglobinemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult or pediatric patients diagnosed with acquired methemoglobinemia and receiving treatment with ProvayBlue® (methylene blue 0.5%) as per the treating physician's diagnosis and the acute care facility's standard of care
* Those acquired methemoglobinemia patients whose diagnosis is aided by measurement of methemoglobin and whose ongoing treatment is guided by re-measurement of methemoglobin ~1h post-treatment with ProvayBlue® in accordance with the US FDA Label prescribing information

Exclusion Criteria:

* Refusal of consent (in those subjects approached for consent where required by local institutional procedures)
* Treatment of methemoglobinemia with another methylene blue product

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present in hospital / urgent care setting diagnosed with acquired methemoglobinemia.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Reduction of Methemoglobin 1h after Administration of ProvayBlue | 1h post-treatment
  Level of methemoglobin 1h after administration of ProvayBlue for treatment of acquired methemoglobinemia compared to pre-treatment level of methemoglobin.

SECONDARY OUTCOMES:
Time to Normalization of Respiratory Rate | Index Hospitalization
  Time to normalization of respiratory rate after administration of ProvayBlue for treatment of acquired methemoglobinemia.
Time to Normalization of Heart Rate | Index Hospitalization
  Time to normalization of heart rate after administration of ProvayBlue for treatment of acquired methemoglobinemia.
Time to Normalization of Blood Pressure | Index Hospitalization
  Time to normalization of blood pressure after administration of ProvayBlue for treatment of acquired methemoglobinemia.
Prevalence and Nature of Adverse Events | Within 10 days of Treatment
  Prevalence and nature of any adverse events occurring within 10 days of the administration of ProvayBlue

OTHER OUTCOMES:
Prevalence by Agent | Index Hospitalization
  Prevalence of acquired methemoglobinemia cases by suspected causal agent
Resolution of Symptoms | Index Hospitalization
  Resolution of methemoglobinemia-related symptoms during the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Charles V Pollack, MD, Principal Investigator — Hospital Quality Foundation
Locations (32):
- United States (32):
  - Cedars Sinai, Los Angeles, California
  - UC Davis Health, Sacramento, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Palmetto General, Palm Beach Gardens, Florida
  - Tampa General, Tampa, Florida
  - IU Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Health System, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Partners Healthcare; Brigham and Women's, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St John Medical Center, Detroit, Michigan
  - HealthPartners Regions, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Methodist, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Mercy Health, Youngstown, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin